CLINICAL TRIAL: NCT04069234
Title: 30-d Rand, Eval-blind, Controlled, Multi-centre, Parallel, ph III Study to Evaluate Effect of a Low Maint Dose Ticagrelor Regimen vs Standard Dose Clopidogrel on Coronary Flow Reserve in DM Patients With Impaired Microvascular Function Without Prior MI or Stroke Undergoing ePCI.
Brief Title: Study in Diabetes Mellitus Patients Without Prior Myocardial Infarction or Stroke Undergoing Elective Percutaneous Coronary Intervention.
Acronym: AUGEAS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decided to stop the study due to commercial reasons.
Sponsor: Region Skane (Other)
Collaborators: IHF GmbH - Institut für Herzinfarktforschung (Other); Hippocrates Research (Other); IRW consulting AB (Unknown); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-04160
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus; Microvascular Coronary Artery Disease
Keywords: myocardial infarction; percutaneous coronary invervention; coronary flow velocity reserve (CFR)
MeSH Terms: conditions — Diabetes Mellitus; Myocardial Infarction | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ticagrelor (Experimental): ticagrelor 60mg BID for 30 Days and ASA 75 - 150 mg once daily
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): clopidogrel 75mg OD for 30 Days and ASA 75 - 150 mg once daily
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — ticagrelor 60 mg BID for 30 days
  Arms: Ticagrelor
Drug: Clopidogrel — clopidogrel 75mg OD for 30 Days
  Arms: Clopidogrel

SUMMARY:
This study is designed to test the hypothesis that ticagrelor is superior to clopidogrel, in improving coronary microvascular function, as measured by coronary flow reserve (CFR) in patients with T2DM at high risk of cardiovascular (CV) events undergoing elective PCI.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) can be divided into macrovascular and microvascular disease, both different manifestations of atherosclerosis. Macrovascular CAD, i.e. obstructive CAD of epicardial coronary arteries have traditionally been the focus of CAD treatment. Microvascular circulation, on the other hand, consists of arterioles (diameter <100 μm) within myocardium and abnormalities in this arterial bed may also impair myocardial perfusion and result in ischaemia. An indication of microvascular disease can be achieved with coronary flow reserve (CFR) which is an integrated measure of flow through both large epicardial arteries and coronary microcirculation. CFR measurement is the ratio of resting coronary artery mean diastolic flow velocity in comparison to hyperaemic coronary artery mean diastolic flow velocity, where hyperaemia is often induced with pharmacologic agent such as adenosine infusion. CFR of the left anterior descending (LAD) coronary artery during pharmacologic stress echocardiography has been found to provide effective prognostic information in patients with known or suspected CAD. This seems evident across patient populations, such as those with diabetes or chronic kidney disease, or older age. Particularly, a CFR <2.0 has been associated with markedly increased cardiovascular (CV) risk in an unselected patient population.

Ticagrelor primary mode of action is as a direct acting reversibly binding P2Y12 antagonist inhibiting ADP-induced platelet activation. However, ticagrelor has also been shown to increase extracellular adenosine concentration by inhibition of the equilibrative nucleoside transporter 1 (ENT1). Adenosine has been described to have a number of physiological effects including vasodilation, anti-inflammation, anti-platelet and cardioprotective effects and ticagrelor has been shown to enhance many of these adenosine-induced effects in animal models and in man. These adenosine-mediated effects may be beneficial to CAD patients and potentially impact coronary microvascular function and contribute to the clinical profile of ticagrelor. So far only one study has explored ticagrelor effect on coronary microvascular function. They showed, by using rubidium 82 positron emission tomography/computed tomography, that ticagrelor could improve local CFR compared to clopidogrel in CAD patients specifically in those regions that before treatment had impaired CFR (<2.5). CFR has been shown to be a strong independent predictor in diabetic patients with suspected coronary disease for future coronary events and survival.

The ongoing THEMIS study is designed to test the hypothesis that ticagrelor is superior to placebo, in prevention of major CV events, as measured by time to first event of the composite of CV death, MI, or stroke in patients with T2DM at high risk of CV events.

Patients undergoing elective PCI are excluded from the THEMIS study as these patients are treated with clopidogrel plus aspirin. The current study is designed to fill this data gap by generating clinically meaningful data with ticagrelor in THEMIS-like patients undergoing elective PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Men or women ≥18 years of age
3. Diagnosed with T2DM defined as treatment with ongoing glucose lowering drug (oral medications and/or insulin) for at least 1 month
4. Presence of CAD undergoing elective PCI
5. Impaired coronary microvascular function post PCI as defined by a CFR ≤2.5 (as per local reading)
6. TIMI 3 flow post PCI

Exclusion Criteria:

1. Previous MI defined as a documented hospitalization with a final diagnosis of spontaneous MI (with the exception of definite secondary MI [e.g., due to coronary revascularization procedure, profound hypotension, hypertensive emergency, tachycardia, or profound anemia]).
2. Previous stroke (transient ischemic attack [TIA] is not included in the stroke definition)
3. Use of an intravenous antiplatelet therapy (i.e., cangrelor or GPI) during PCI
4. On treatment with clopidogrel, prasugrel, or ticagrelor due to a prior acute major CV event (MI or stroke) (on treatment with clopidogrel due to prior vascular intervention not secondary to a major CV event is allowed)
5. Planned use of aspirin treatment at doses >150 mg od
6. Anticipated concomitant oral or intravenous therapy with strong cytochrome P450 3A4 (CYP3A4) inhibitors or CYP3A4 substrates with narrow therapeutic indices that cannot be stopped for the course of the study:

   1. Strong CYP3A4 inhibitors: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin (but not erythromycin or azithromycin), nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir
   2. CYP3A4 substrates with narrow therapeutic index: quinidine, simvastatin at doses >40 mg daily or lovastatin at doses >40 mg daily
7. Hypersensitivity to ticagrelor or any of its excipients
8. Need for chronic oral anticoagulant therapy or chronic low-molecular-weight heparin
9. Patients with known bleeding diathesis or coagulation disorder
10. History of intracerebral bleed at any time, gastrointestinal (GI) bleed within the past 6 months prior to randomization, or major surgery within 30 days prior to randomization
11. Increased risk of bradycardic events (e.g., known sick sinus syndrome, second or third-degree AV block or previous documented syncope suspected to be due to bradycardia) unless treated with a pacemaker
12. Known severe liver disease (e.g., ascites and/or clinical signs of coagulopathy)
13. Renal failure requiring dialysis
14. Known platelet count <145 x109 platelets/L
15. Known hemoglobin <9 g/dL
16. Women of child-bearing potential (WOCBP)*, who are not willing to use a method of contraception that is considered highly reliable** per CTFG (Clinical Trial Facilitation Group), OR who have a positive pregnancy test at enrolment or randomization OR women who are breast-feeding
17. Inability of the patient to understand and/or comply with study procedures and/or follow up, in the opinion of the investigator, OR any conditions that, in the opinion of the investigator, may render the patient unable to complete the study
18. Life expectancy of less than 6 month based on investigator's judgement
19. Participation in another clinical study with an investigational (defined as non-approved) product, if taken within five half-lives or 28 days prior to the first administration of the trial medication, whichever is longer
20. Previous randomization in the present study
21. Severe asthma
22. Hypersensitivity to adenosine or mannitol
23. Long QT syndrome
24. Chronic obstructive lung disease, with evidence of bronchospasm
25. Severe low blood pressure
26. Unstable angina pectoris
27. Severe heart failure
28. Hypovolemia
29. Treatment with dipyradimol
30. Increased intracranial pressure * fertile, following menarche until becoming post-menopausal, unless permanently sterile (permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy) ** estrogen/progestogen or progestogen (oral, intravaginal or transdermal administration); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2021-10-15 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Coronary Flow Velocity Reserve (CFR) | 30+/- 3 days after randomization
  Difference in mean of individual absolute change from baseline to 30 days in Coronary Flow Velocity Reserve (CFR) in the mid-distal segment of the left anterior descending (LAD) coronary artery under adenosine infusion measured by Transthoracic Doppler Echocardiography (TDE) between the two arms

SECONDARY OUTCOMES:
Coronary flow parameter-LAD hyperemic mean diastolic flow velocity | 30+/- 3 days after randomization
  Difference in mean of individual absolute change from baseline at 30 days in:
  - LAD hyperemic mean diastolic flow velocity
Coronary flow parameter-LAD resting mean diastolic flow velocity | 30+/- 3 days after randomization
  Difference in mean of individual absolute change from baseline at 30 days
  - LAD resting mean diastolic flow velocity